CLINICAL TRIAL: NCT03573115
Title: Multimodal Optical Imaging for Pretreatment Evaluation for Cutaneous Microparticle Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Collaborators: Sebacia, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Clinical Professor, Consultant in Dermatology (DMSc, PhD, MD), Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EudraCT: 2017-002975-25
Record Dates: First submitted 2018-05-02; First posted 2018-06-29 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Acne Vulgaris; Microparticles
Keywords: Optical Coherence Tomography; Reflectance Confocal Microscopy; Gold microparticles; Adapalene; Benzoyl Peroxide
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acne patients (Experimental)
  Interventions: Drug: Adapalene-Benzoyl Peroxide Gel 0.1-2.5%

INTERVENTIONS:
Drug: Adapalene-Benzoyl Peroxide Gel 0.1-2.5% — Topical gold microparticles (SEB-250) are delivered to two facial areas at baseline, patients are then prescribed a topical Adapalene-Benzoyl Peroxide Gel 0.1-2.5% for 6 weeks followed by a new exposure to gold microparticles (SEB-250)
  Other Names: Seb-250

SUMMARY:
The purpose of this study is to investigate how pretreatment with a topical medication for acne affects application and delivery of gold microparticles to the skin in acne patients. In addition, the investigators want to investigate the biodistribution of gold microparticles in pretreated skin and compare this with the biodistribution of untreated skin using the non-invasive imaging techniques optical coherence tomography and reflectance confocal microscopy

DETAILED DESCRIPTION:
Epiduo is a prescription gel that combines adapalene and benzoyl peroxide, two active substances for the external treatment of acne. Adapalene is a substance that resembles A-vitamin acid, which dissolves and prevents clog formation in the sebaceous glands. Benzoyl peroxide works by reducing the amount of bacteria while dissolving the clogs in the sebaceous glands. Epiduo is the only antibiotic-free combination for the treatment of acne.

Reflectance Confocal Microscopy (RCM) and Optical Coherence Tomography (OCT) are non-invasive imaging technologies allowing for imaging of the upper skin layers. Gold microparticles have been shown to have a contrast effect on the images. In addition to the contrast effect on images, gold microparticles have proven to be effective in the treatment of skin disease acne. The treatment with gold microparticles uses a combination of the gold microparticles and a laser. The microparticles consist of very small particles of silica, surrounded by a shell of gold. These two components of the microparticles are selected from their way of absorbing light from a laser. The particles absorb the light from the laser and are thus heated. The surrounding skin can not absorb the light and therefore will maintain its normal temperature.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical diagnosis of acne vulgaris, IGA score 1-3
2. 18-45 years of age at baseline
3. Legally competent, able to give verbal and written consent
4. Communicate in Danish verbally as well as in writing
5. Fitzpatrick skin phototype I-III
6. Subjects in good general health, willing to participate and able to give informed consent, and can comply with protocol requirements
7. Female subjects of childbearing potential (1) must be confirmed not pregnant by a negative urine pregnancy test prior to trial treatment
8. Female subjects must use one of following contraceptive techniques to be included in the study: intrauterine device (IUD) or hormonal contraception (birth control pills, birth control patch, birth control vaginal ring, birth control shot or birth control implant) (1) Female subjects are considered of childbearing potential unless they have been hysterectomized

Exclusion Criteria:

1. Subjects with a known allergy to gold microparticles or Epiduo®
2. Individuals with other skin disease than acne or skin lesions in the area of research interest
3. Subjects with tattoo in the treatment area which may interfere with or confound evaluation of the study
4. Subjects with moderate-severe to severe acne (IGA 4-5 and those presenting with either cysts or nodules) requiring continuation of systemic treatment during the study period
5. Subjects with a history of keloids which is deemed clinically relevant in the opinion of the investigator
6. Subjects with active skin disease or excessive scarring that, in the opinion of the investigator, would impact the ability to administer the gold microparticles or use of OCT/RCM in the areas
7. Pregnant and lactating women
8. Subjects who have received investigational drugs or were treated with investigational devices within 30 days prior to baseline
9. Treatment with oral retinoid 3 months prior to baseline
10. Treatment with systemic antibiotics 4 weeks prior to baseline
11. Topical retinoids, topical antibiotics or topical products with benzoyl peroxide 4 weeks prior to baseline

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in gold microparticle delivery after 6 weeks of pretreatment evaluated by RCM | baseline and after 6 weeks of study
  Quantitative evaluation of fraction of follicles with gold microparticles at baseline and after 6 weeks of study. Change in fraction of follicles with gold will be assessed.
Change in gold microparticle delivery after 6 weeks of pretreatment evaluated by OCT | baseline and after 6 weeks of study
  Quantitative evaluation of depth of gold in hair follicles at baseline and after 6 weeks of pretreatment, measured in um. Change in depth will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Department of Dermatology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided